CLINICAL TRIAL: NCT02909751
Title: Tocotrienol in Combination With Neoadjuvant Chemotherapy for Women With Breast Cancer
Acronym: NeoToc
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NeoToc
Record Dates: First submitted 2016-09-16; First posted 2016-09-21 (Estimated); Last update posted 2021-05-20 (Actual); Status verified 2021-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Epirubicin; Cyclophosphamide; Docetaxel; Paclitaxel; Trastuzumab; pertuzumab; Tocotrienols

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Neoadjuvant chemotherapy (Active Comparator): HER2 negative:
  Four cycles of 3-weekly epirubicin 90 mg/m2 iv and cyclophosphamid 600 mg/m2 iv followed by Four cycles of taxane, i.e. 3-weekly docetaxel 100 mg/m2 iv or weekly paclitaxel 80 mg/m2 iv
  HER2 positive:
  Four cycles of taxane, i.e. 3-weekly docetaxel 100 mg/m2 iv or weekly paclitaxel 80 mg/m2 iv + 3-weekly trastuzumab (8 mg/kg iv saturation, then 6 mg/kg iv) and possibly pertuzumab (840 mg saturation, then 420 mg iv) followed by Four cycles of 3-weekly epirubicin 90 mg/m2 iv and cyclophosphamid 600 mg/m2 iv
  Interventions: Drug: Epirubicin 90 mg/m2 iv; Drug: Cyclophosphamide 600 mg/m2 iv; Drug: Docetaxel 100 mg/m2 iv OR paclitaxel 80 mg/m2 iv; Drug: Trastuzumab 8 mg/kg iv saturation, then 6 mg/kg iv (HER2 positive patients only); Drug: Pertuzumab 840 mg iv saturation, then 420 mg iv (selected HER2 positive patients only)
- Neoadjuvant chemotherapy + tocotrienol (Experimental): HER2 negative:
  Four cycles of 3-weekly epirubicin 90 mg/m2 iv and cyclophosphamid 600 mg/m2 iv followed by Four cycles of taxane, i.e. 3-weekly docetaxel 100 mg/m2 iv or weekly paclitaxel 80 mg/m2 iv.
  Daily: Tocotrienol 300 mg x 3
  HER2 positive:
  Four cycles of taxane, i.e. 3-weekly docetaxel 100 mg/m2 iv or weekly paclitaxel 80 mg/m2 iv + 3-weekly trastuzumab (8 mg/kg iv saturation, then 6 mg/kg iv) and possibly pertuzumab (840 mg saturation, then 420 mg iv) followed by Four cycles of 3-weekly epirubicin 90 mg/m2 iv and cyclophosphamid 600 mg/m2 iv.
  Daily: Tocotrienol 300 mg x 3
  Interventions: Drug: Epirubicin 90 mg/m2 iv; Drug: Cyclophosphamide 600 mg/m2 iv; Drug: Docetaxel 100 mg/m2 iv OR paclitaxel 80 mg/m2 iv; Drug: Trastuzumab 8 mg/kg iv saturation, then 6 mg/kg iv (HER2 positive patients only); Drug: Pertuzumab 840 mg iv saturation, then 420 mg iv (selected HER2 positive patients only); Dietary Supplement: Tocotrienol 300 mg x 3 daily

INTERVENTIONS:
Drug: Epirubicin 90 mg/m2 iv — Max. 3 months
Drug: Cyclophosphamide 600 mg/m2 iv — Max. 3 months
Drug: Docetaxel 100 mg/m2 iv OR paclitaxel 80 mg/m2 iv — Max. 3 months
Drug: Trastuzumab 8 mg/kg iv saturation, then 6 mg/kg iv (HER2 positive patients only) — Max. 3 months.
Drug: Pertuzumab 840 mg iv saturation, then 420 mg iv (selected HER2 positive patients only) — Max. 3 months
Dietary Supplement: Tocotrienol 300 mg x 3 daily — Max. 6 months
  Arms: Neoadjuvant chemotherapy + tocotrienol

SUMMARY:
The purpose of this study is to investigate whether tocotrienol can improve the effect and reduce the side effects of standard chemotherapy before operation for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Women with histologically verified breast cancer (adenocarcinoma)
* Age ≥ 18 years.
* Neoadjuvant treatment indicated according to departmental guidelines
* PS 0-2 and suited for surgery.
* Normal heart function, LVEF ≥ 50% by MUGA/ECHO in patients receiving neoadjuvant trastuzumab
* Normal bone marrow function: Hemoglobin ≥ 6 mmol/l; ANC ≥ 1.5x10^9/l; Thrombocytes ≥ 100x10^9/l.
* Normal liver function: Bilirubin ≤ 1.5 x upper level of normal, ALAT ≤ 2.5 x upper level of normal, BASP ≤ 2.5 x upper level of normal.
* Normal kidney function: Creatinine ≤ upper level of normal. In case of increased creatinine, measured/calculated GFR must be ≥ 50 ml/min.
* Fertile women must present a negative pregnancy test and use a safe contraceptive during and 3 months after the treatment. Intrauterine device without hormone is considered safe.
* Written and orally informed consent

Exclusion Criteria:

* Bilateral breast cancer or suspected dissemination. Verified by bilateral mammography, bone scintigraphy, chest and abdomen CT, and PET-CT.
* Pregnant and breastfeeding women
* Mental or social conditions that will prevent treatment or follow-up
* Other simultaneous experimental treatment
* Immunosuppressive treatment (other than prednisolone during neoadjuvant chemotherapy)
* Vitamin or nutritional supplements (other than multivitamin tablet and calcium tablet with vitamin D)
* Active or latent viral/bacterial infection
* Rheumatoid arthritis or other autoimmune disease
* Other malignant disease within the past 5 years excl. non-melanoma cancer of the skin and carcinoma in situ cervicis uteri.
* Previous treatment with docetaxel, paclitaxel, epirubicin, cyclophosphamide, trastuzumab, pertuzumab or tocotrienol
* Hypersensitivity to any of the active or auxiliary substances

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2019-01-21 (Actual); Study Completion 2019-01-21 (Actual)

PRIMARY OUTCOMES:
Pathological complete response | 26 weeks from date of inclusion

SECONDARY OUTCOMES:
Correlation of changes in NK-cells with pathological complete response | 26 weeks from date of inclusion
Correlation of changes in ctDNA with pathological complete response | 26 weeks from date of inclusion
Number of patients with grade 3-4 side effects | 29 weeks from date of inclusion

CONTACTS AND LOCATIONS:
Overall Officials: Erik H Jakobsen, MD, Study Chair — Vejle Hospital
Locations (1):
- Vejle hospital, Department of Oncology, Vejle, Denmark